CLINICAL TRIAL: NCT00764660
Title: A Prospective, Double-Blind, Placebo-Controlled Trial Investigating the Efficacy and Safety of SCH 900435 (Org 25935) in Relapse Prevention in Subjects With Alcohol Dependence.
Brief Title: Trial Investigating the Efficacy and Safety of SCH 900435 (Org 25935) in Relapse Prevention in Participants With Alcohol Dependence (P05718)
Acronym: OD-H
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on the outcome of a planned interim analysis, the study was stopped early due to futility.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05718; 2008-005318-35 (EudraCT Number); 172009 (Other: Organon Protocol Number); MK-8435-003 (Other: Merck Protocol Number)
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — N-methyl-N-(6-methoxy-1-phenyl-1,2,3,4-tetrahydronaphthalen-2-ylmethyl)aminomethylcarboxylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCH 900435 (Experimental): Participants received SCH 900435 12 mg (as three SCH 900435 4 mg tablets) by mouth twice daily for 12 weeks.
  Interventions: Drug: SCH 900435
- Placebo (Placebo Comparator): Participants received matching placebo tablets by mouth twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCH 900435 — tablets
  Other Names: Org 25935; MK-8435
  Arms: SCH 900435
Drug: Placebo — tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effects of SCH 900435 (Org 25935, MK-8435) on heavy drinking, safety and tolerability of SCH 900435 in participants with alcohol dependence.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent after the scope and nature of the investigation, have been explained to the participant before screening;
* Diagnosis of alcohol dependence - meeting at least 5 out of 7 criteria according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) specifier; one of which should be criterion 1 (tolerance) or 2 (withdrawal);
* Primary complaints according to Mini-International Neuropsychiatric Interview (MINI) should be alcohol problems;
* Participants must have gone through a detoxification program, have a clearly stated desire to stay abstinent and present at baseline with the following: be alcohol abstinent for at least 3 days, benzodiazepine free for at least 3 days, and a Clinical Institute Withdrawal Assessment (CIWA) score <10;
* Age 18-65 years at screening;
* Males, or females who are not of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year) or who are non-pregnant, non-lactating and using a medically accepted method of contraception; these include condoms with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed intrauterine device (IUD), and hormonal contraceptives;
* Body Mass Index (BMI) >16 kg/m^2;
* Breath alcohol concentration < 0.02% (at screening and baseline)

Exclusion Criteria:

* Participants requiring pharmacological treatment for a primary diagnosis of major depressive disorder, anxiety, panic disorder or social phobia;
* Participants with psychotic disorders (according to MINI);
* Participants with a medium or high suicidality risk (as assessed by MINI)
* Active substance abuse (resulting in either physical or mental damage as defined by International Statistical Classification of Diseases and Related Health Problems, 10th revision [ICD10] or dependence other than alcohol (excluding nicotine) within 12 months prior to screening, e.g. cannabis, benzodiazepine, amphetamines, chlo(r)methiazole, opiates, cocaine, hallucinogens or other substances;
* Use of one of the following drugs during the last 14 days prior to screening: cannabis, amphetamines, opiates, cocaine, hallucinogens;
* Use of any medication that can have an effect on alcohol consumption within 30 days of study initiation, including naltrexone, acamprosate, disulfiram, ondansetron, topiramate, selective serotonin reuptake inhibitors (SSRIs), mirtazapine, varencicline, gabapentin, levetiracetam;
* A clinically relevant visual disturbance, such as cataract, color blindness, macular degeneration, glaucoma or retinal disease;
* Untreated or uncompensated clinically significant renal, endocrine, hepatic, respiratory, cardiovascular, hematological, immunological or cerebrovascular disease, malignancy, or other chronic and/or degenerative process at screening;
* Any clinically meaningful abnormal laboratory, vital sign, physical examination or electrocardiogram (ECG) finding which, in the opinion of the investigator, may interfere with the interpretation of safety or efficacy evaluations;
* QTc interval (Fridericia corrected) at screening >450 ms (male), >470 ms (female);
* Serious neuropsychiatric condition that can impair judgment or cognitive function (including dementia or amnestic disorder) to an extent that providing informed consent or complying with treatment is precluded;
* History or present evidence of epileptic disorders or withdrawal seizures;
* History of substance withdrawal delirium;
* Breast-feeding woman, or a positive result of urine pregnancy test (at screening), or plan to become pregnant during the course of the trial (females only);
* Pending legal charges with the potential for incarceration, probation, or parole;
* Homelessness (less than 2 months stable residence);
* Participation in a clinical trial during the 3 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2009-02-13 (Actual); Primary Completion 2010-05-28 (Actual); Study Completion 2010-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] de Bejczy A, Nations KR, Szegedi A, Schoemaker J, Ruwe F, Soderpalm B. Efficacy and safety of the glycine transporter-1 inhibitor org 25935 for the prevention of relapse in alcohol-dependent patients: a randomized, double-blind, placebo-controlled trial. Alcohol Clin Exp Res. 2014 Sep;38(9):2427-35. doi: 10.1111/acer.12501. PMID 25257291

RESULTS

PARTICIPANT FLOW:
Groups:
- SCH 900435 12 mg: Participants received SCH 900435 12 mg (as three SCH 900435 4 mg tablets) by mouth twice daily for 12 weeks.
Period: Overall Study
Arm/Group | SCH 900435 12 mg | Placebo
Started | 75 | 66
Completed | 53 | 55
Not Completed | 22 | 11
Not completed — Adverse Event | 6 | 3
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Noncompliance With Protocol | 5 | 1
Not completed — Did Not Meet Protocol Eligibility | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCH 900435 12 mg | Placebo | Total
Number analyzed (Participants) | 75 | 66 | 141
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.5 (10.3) | 50.3 (9.3) | 49.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 55 | 49 | 104

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Heavy Drinking Days
Description: Percentage of heavy drinking days was defined as days with ≥5 standard drinks for men and ≥4 standard drinks for women assessed by Alcohol Timeline Follow Back (TLFB) method. The Alcohol TLFB is a drinking assessment method that obtains estimates of daily drinking by means of an interview between investigator and participant. The TLFB assesses recent drinking behavior. On the TLFB, clients retrospectively estimate their daily alcohol consumption in standard drinks over a time period prior to the interview, and thus the measure provides quantitative estimates of alcohol use.
  A drink is standardized to an equivalent to 25-30 cL of beer or wine coolers (5% alcohol), 12-15 cL of table wine (11-14% alcohol) and 4-6 cL of hard liquor/spirits (35-40% alcohol).
  Percentage was calculated based on number of heavy drinking days divided by total number of days in the given 2-week interval.
Time Frame: 12 weeks
Population: The modified Intent-to-Treat (mITT) population consisted of all participants from the All-Participants-Treated (APT) population who had at least post randomization efficacy data for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Days
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 74 | 65
Percentage of Days | 18.7 [14.5 to 23.0] | 16.3 [11.8 to 20.8]
Statistical Analysis 1: Comparison: SCH 900435 12 mg vs Placebo; Test type: Superiority or Other; p = 0.41, Repeated Measures Model; Difference in LS Means = 2.4, 95% CI 2-sided [-3.4 to 8.2] — Repeated Measures Model with factors for treatment, pooled centers, assessment and assessment by treatment interaction

2. Secondary Outcome: Number of Drinks Per Drinking Day
Description: The amount of drinking was defined as drinks per drinking day (TLFB). Drinking day is a day on which an alcoholic drink is consumed, with 'day' being defined as the period between waking up and going to sleep; the end of a day may have crossed the time point of midnight.
Time Frame: 12 weeks
Population: The mITT population consisted of all participants from the APT population who had at least post randomization efficacy data for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Drinks
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 49 | 47
Drinks | 10.9 [8.2 to 13.5] | 12.8 [9.9 to 15.6]
Statistical Analysis 1: Comparison: SCH 900435 12 mg vs Placebo; Test type: Superiority or Other; p = 0.30, Repeated Measures Model; Difference in Least Squares (LS) Means = -1.9, 95% CI 2-sided [-5.5 to 1.7] — Repeated Measures Model with factors for treatment, pooled centers, assessment and assessment by treatment interaction

3. Secondary Outcome: Number of Relapses Into Heavy Drinking
Description: An alcohol relapse was defined as either a daily alcohol intake of 5 or more drinks for males and 4 or more drinks for females or an overall consumption of 14 drinks or more per week during at least 4 weeks (TLFB).
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Relapses
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 74 | 65
Relapses | 4.65 (6.24) | 4.52 (5.27)
Statistical Analysis 1: Comparison: SCH 900435 12 mg vs Placebo; Test type: Superiority or Other; p = 0.52, Chi-squared; Zero Inflated Negative Binomial (ZINB) Distribution with terms for treatment and region; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.57 to 1.33]

4. Secondary Outcome: Number of Lapses Into Any Drinking
Description: An alcohol lapse was defined as any episode of alcohol consumption not classified as a relapse (TLFB).
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Lapses
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 74 | 65
Lapses | 5.59 (6.33) [0.31 to 4.86] | 6.37 (6.49) [0.24 to 4.73]
Statistical Analysis 1: Comparison: SCH 900435 12 mg vs Placebo; Test type: Superiority or Other; p = 0.81, Chi-squared; ZINB Distribution with terms for treatment and region; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.71 to 1.31]

5. Secondary Outcome: Time to First Relapse Into Drinking
Description: Time to relapse was defined as the time to first relapse into heavy drinking (TLFB). A Hazard Ratio (SCH 900435/Placebo) of <1 means that SCH 900435 has a lower risk of relapsing as compared to Placebo.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 74 | 65
Days | 37.1 (35.5) | 41.6 (36.3)
Statistical Analysis 1: Comparison: SCH 900435 12 mg vs Placebo; Test type: Superiority or Other; p = 0.26, Kaplan-Meier — Model with factors treatment and pooled centers as stratum; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.81 to 2.12]

6. Secondary Outcome: Percentage of Abstinent Days
Description: Percentage of abstinent days is the percentage of study days in which participants remained abstinent during the treatment period.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Days
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 74 | 65
Percentage of Days | 70.5 [64.9 to 76.2] | 72.6 [66.6 to 78.6]
Statistical Analysis 1: Comparison: SCH 900435 12 mg vs Placebo; Test type: Superiority or Other; p = 0.59, Repeated Measures Model; Repeated Measures Model with factors for treatment, pooled centers, assessment and assessment by treatment interaction; Difference in LS Means = -2.1, 95% CI 2-sided [-9.9 to 5.7]

7. Secondary Outcome: Percentage of Participants With Complete Abstinence
Description: Percentage of total abstinence is the percentage of participants who remained abstinent during the entire treatment period.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 74 | 65
Percentage of Participants | 33.8 [64.9 to 76.2] | 27.7 [66.6 to 78.6]
Statistical Analysis 1: Comparison: SCH 900435 12 mg vs Placebo; Test type: Superiority or Other; p = 0.34, Regression, Logistic; An Odds Ratio (SCH 900435/Placebo) >1 means SCH 900435 has a higher probability of achieving complete abstinence; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.65 to 3.43]

8. Secondary Outcome: Global Functioning: Clinical Global Impression (CGI) - Severity of Illness
Description: The CGI scale is a standardized tool used by investigators to rate the severity of illness, taking into account the participant's clinical condition and the severity of side effects. The CGI scores could range from 1 to 7, with a lower score reflecting a better outcome.
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 34 | 38
Score on a Scale | 2.7 (1.3) | 2.7 (1.4)

9. Secondary Outcome: Global Functioning: CGI - Therapeutic Effect
Description: The CGI scale is a standardized tool used by investigators to rate the efficacy of study drug (therapeutic effect), taking into account the participant's clinical condition and the severity of side effects. The CGI scores could range from 1 to 7, with a lower score reflecting a better outcome.
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 34 | 38
Score on a Scale | 2.1 (1.2) | 2.0 (1.0)

10. Secondary Outcome: Change From Baseline in Craving Visual Analog Scale (VAS) Score
Description: Rating of craving is included to assess a potential relationship between treatment and craving severity. Participants were asked to answer the question: "Over the past week, what has your desire or craving for an alcoholic beverage been at the time of day that you usually drink?" The 100 mm line of the VAS was anchored on the left by "No desire at all" and on the right by "Extreme desire". Participants marked a spot on the line where they felt their craving severity fit best. Craving VAS scores could range from 0 to 100, with a lower VAS score reflecting a better outcome.
Time Frame: Baseline and Day 84
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 36 | 39
Score on a Scale | -3.56 [-10.53 to 3.41] | -6.44 [-13.25 to 0.38]
Statistical Analysis 1: Comparison: SCH 900435 12 mg vs Placebo; Test type: Superiority or Other; p = 0.54, Contrained Longitudinal Data Analysis; Difference in LS Means = 2.88, 95% CI 2-sided [-6.30 to 12.06] — Constrained Longitudinal Data Analysis (cLDA) Model with terms for treatment, pooled centers, assessment by treatment interaction

11. Secondary Outcome: Change From Baseline in Motivation VAS Score
Description: Participants were asked to answer the question: "Over the past week, how motivated were you to stay alcohol abstinent?" The 100 mm line of the VAS was anchored on the left by "No motivation at all" and on the right by "Extremely motivated". Motivation VAS scores could range from 0 to 100, with a higher score reflecting a better outcome.
Time Frame: Baseline and Day 84
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 36 | 39
Score on a Scale | -8.09 [-14.85 to -1.33] | -4.99 [-11.66 to 1.68]
Statistical Analysis 1: Comparison: SCH 900435 12 mg vs Placebo; Test type: Superiority or Other; p = 0.51, cLDA Model; Difference in LS Means = -3.10, 95% CI 2-sided [-12.35 to 6.15] — cLDA Model with terms for treatment, pooled centers, assessment by treatment interaction

12. Secondary Outcome: Change From Baseline in Mood VAS Score
Description: Participants were asked to answer the question: "Over the past week, how did you feel?" The 100 mm line of the VAS was anchored on the left by "Extremely bad" and on the right by "Extremely good". Mood VAS scores could range from 0 to 100, with a higher VAS score reflecting a better outcome.
Time Frame: Baseline and Day 84
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 36 | 39
Score on a Scale | -5.29 [-12.01 to 1.42] | 3.88 [-2.74 to 10.49]
Statistical Analysis 1: Comparison: SCH 900435 12 mg vs Placebo; Test type: Superiority or Other; p = 0.05, cLDA Model; Difference in LS Means = -9.17, 95% CI 2-sided [-18.27 to -0.07] — cLDA Model with terms for treatment, pooled centers, assessment by treatment interaction

13. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not related to the study drug.
Time Frame: Up to 16 weeks
Population: The All-Participants-Treated (APT) population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 75 | 66
Participants | 65 | 53

14. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 13
Time Frame: Up to 12 weeks
Population: The APT population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | SCH 900435 12 mg | Placebo
Number analyzed (Participants) | 75 | 66
Participants | 6 | 3

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Description: The APT population consisted of all participants who received at least one dose of study drug.
Arm/Group | SCH 900435 12 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 10/75 | 11/66
Other Adverse Events (participants affected / at risk) | 53/75 | 43/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 900435 12 mg (N=75) | Placebo (N=66)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEPATITIS CHOLESTATIC (Hepatobiliary disorders) | 1 (1) | 0 (0)
ABSCESS SWEAT GLAND (Infections and infestations) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 1 (1) | 0 (0)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BLOOD PRESSURE ABNORMAL (Investigations) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1) | 0 (0)
GRAND MAL CONVULSION (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
ALCOHOLISM (Psychiatric disorders) | 0 (0) | 1 (1)
DRUG WITHDRAWAL MAINTENANCE THERAPY (Surgical and medical procedures) | 3 (3) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 900435 12 mg (N=75) | Placebo (N=66)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
PHOTOPHOBIA (Eye disorders) | 9 (9) | 1 (1)
PHOTOPSIA (Eye disorders) | 6 (7) | 2 (2)
VISION BLURRED (Eye disorders) | 5 (6) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 7 (9) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 6 (9) | 7 (8)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 5 (7) | 6 (7)
FATIGUE (General disorders) | 19 (22) | 9 (9)
INFLUENZA (Infections and infestations) | 6 (6) | 7 (7)
NASOPHARYNGITIS (Infections and infestations) | 11 (18) | 18 (21)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (7)
BALANCE DISORDER (Nervous system disorders) | 5 (6) | 0 (0)
DIZZINESS (Nervous system disorders) | 15 (19) | 3 (5)
HEADACHE (Nervous system disorders) | 13 (23) | 15 (17)
TUNNEL VISION (Nervous system disorders) | 4 (4) | 0 (0)
VISUAL FIELD DEFECT (Nervous system disorders) | 4 (5) | 1 (2)
INSOMNIA (Psychiatric disorders) | 6 (6) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In case the proposed publication contains reference to an invention owned by Organon or to which Organon otherwise has rights, Organon may request a reasonable suspension of the publication in order to be able to file a patent application protecting such invention.